CLINICAL TRIAL: NCT01926821
Title: The Impact of Sonifilan on the Quality of Life in Patients With Cervical Cancer
Brief Title: Impact of Sonifilan on the Quality of Life in Patients With Cervical Cancer During Radiation or Chemoradiation Therapy
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Jong-Hyeok Kim, Professor, Asan Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SIZO2013
Record Dates: First submitted 2013-08-19; First posted 2013-08-21 (Estimated); Last update posted 2017-05-31 (Actual); Status verified 2017-05

CONDITIONS: Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Sizofiran

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- sonifilan (Experimental): Group who get sonifilan
  Interventions: Drug: Sonifilan
- control (No Intervention): No Sonifilan administered

INTERVENTIONS:
Drug: Sonifilan — Sonifilan inj 20mg Intra muscular injection, twice per week for 8 weeks, total 16 times
  Other Names: sizofiran inj 20mg; Code : XSISO
  Arms: sonifilan

SUMMARY:
The impact of sonifilan on the quality of life in patients with cervical cancer during radiation or chemoradiation therapy

1. Primary endpoint : Quality of life
2. Secondary endpoint : complications related to Sonifilan, treatment effect of Sonifilan

DETAILED DESCRIPTION:
Study design Prospective randomized controlled trial

Study period Protocol registration approval date - may/31/2016

Study drug Sonifilan(Sizofiran)

Study population

1. Cervical cancer FIGO stage IA2-IVA patients will be participated.
2. Squamous cell carcinoma, adenocarcinoma, adenosquamous carcinoma
3. age 20-75 year

Treatment Fron the day of radiation therapy started, Sonifilan 20mg, 1amp IM/week for 8weeks

Concurrent therapy Chemo & radiation therapy

1. Cisplatin 40mg/m2, day 1, 8, 15, 2, 29, 36
2. External whole pelvic irradiation 3000-3500 cGy / 6 fractions in high dose rate

Assessment

1. Pre-study assessment (within 4weeks before participation) a medical history b informed consent c ID number assignment d life quality assessment - fill out EORTC QOQ-C30, CX24, SF-36, FSFI e basic information collect
2. On-study assessment (during study) a complication check b life quality assessment - fill out EORTC QOQ-C30, CX24, SF-36, FSFI

3. Post-study assessment (1week after study finished) a MRI b PAP smear c HPV test d life quality assessment - fill out EORTC QOQ-C30, CX24, SF-36, FSFI

4 Follow-up assessment (every 3 month for 1 year) a Pelvic exam b PAP smear c HPV test d MRI (if needed) e PET (if needed) f life quality assessment - fill out EORTC QOQ-C30, CX24, SF-36, FSFI 93, 6, 12, 24 month after study finished)

ELIGIBILITY:
Inclusion Criteria:

* Cervical cancer FIGO stage IA2 - IVA
* Histologic type : SCC, Adenocarcinoma, Adenosquamous carcinoma
* GOG performance status 0-2

Exclusion Criteria:

* past radiation therapy history
* Neuroendocrine carcinoma
* concurrent other cancer
* uncontrolled medical disease
* ulcerative disease history
* current pregnancy and lactation

Ages: 20 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2013-05; Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Quality of life | 3 year
  life quality assessment by filling out EORTC QOQ-C30, CX24, SF-36, FSFI pre-/on-/post-study

SECONDARY OUTCOMES:
Complications of drug, treatment effects | 3 year

CONTACTS AND LOCATIONS:
Overall Officials: jongHyeok Kim, PhD, Study Chair — Asan Medical Cneter
Locations (1):
- JongHyeokKim, Seoul, South Korea